CLINICAL TRIAL: NCT06538454
Title: Acute and Chronic Effects of Resistance Training Intensity on Cardiovascular Parameters of Postmenopausal Women With Systemic Arterial Hypertension
Brief Title: Effects of Resistance Training Intensity on Cardiovascular Parameters of Hypertensive Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Leonardo da Silva Gonçalves, Principal Investigator, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LOADPMW5065
Record Dates: First submitted 2024-07-29; First posted 2024-08-05 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-08

CONDITIONS: Arterial Hypertension; Postmenopausal; Menorrhagia; Cardiovascular Diseases
Keywords: Resistance training; Intensity; Blood pressure; Heart rate variability; Endothelial function
MeSH Terms: conditions — Hypertension; Menorrhagia; Cardiovascular Diseases | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: The study will be conducted in two stages: one acute and one chronic. In the acute stage, with a crossover design, the subjects will be perform in a random order two resistance training sessions with different intensity. Following this stage, the subjects will be randomized in one of two groups of intensity in a randomized clinical trial design with 10 week of intervention (resistance training).
Who Masked: Investigator
Masking Description: Exercise training studies cannot blind therapists or participants to the intervention or exercise administred. Our study will blind the statistical analysis because we will code the data to avoid knowledge about the intervention performed and who was the participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 80% of 1 repetition maximum (Active Comparator): The recent guideliness suggest a resistance training intensity for this population between 50 and 80% of 1 repetition maximum (1RM), i.e, this group will training in accordance with the recommendations.
  These group will be training with 80% 1RM, performining 8-10 repetitions per set.
  Interventions: Behavioral: Resistance training
- 60% of 1 repetition maximum (Active Comparator): The recent guideliness suggest a resistance training intensity for this population between 50 and 80% of 1 repetition maximum (1RM), i.e, this group will training in accordance with the recommendations.
  These group will be training with 60% 1RM, performining 18-20 repetitions per set.
  Interventions: Behavioral: Resistance training

INTERVENTIONS:
Behavioral: Resistance training — The exercises will be the same in both stages: squat, bench press, stiff, rowing, hip thrust and shoulder press. Futhermore, the rest interval (2 minutes) and the exercise order (alterning upper and lower limbs) also will be the same in the stages.
  In the chronic experiment, the resistance training will be carried for 10 weeks with 2 weekly sessions in alternate days. The sets in both groups will be carried close to muscle failure.
  The difference between groups is the intensity, who reflects the repetition zone. The 80%1RM group will be perform 8-10 repetitions per set, while the 60%1RM group will be perform 18-20 repetitions.
  Other Names: Strength training

SUMMARY:
The goal of this clinical trial is to understand about the effects of resistance training (RT) intensity on cardiovascular parameters in postmenopausal women with systemic arterial hypertension (SAH). The main research questions are:

* Does the intensity of RT impact blood pressure (BP) in postmenopausal women with SAH?
* How does RT intensity affect heart rate (HR) and their variability (HRV), endothelial function (EF), and nitric oxide (NO) biomarker synthesis in this population?
* What are the effects of RT intensity on affectivity and rate of perceived exertion (RPE)?

Researchers will compare two different intensities of RT (60% of the load for 1 repetition maximum [1RM] and 80% of 1RM) to determine their effects on the mentioned cardiovascular and perceptual parameters.

Participants will:

In the acute experiment:

* Perform the same RT session in a crossover design, training with 60% of 1RM in one condition and 80% of 1RM in another condition
* Have BP, HR, and HRV measured before, immediately after, and for one hour post-session
* Report affectivity before each session and at the end, along with RPE

In the chronic experiment:

* Be randomized into two groups: one training with 60% of 1RM and the other with 80% of 1RM
* Undergo a 10-week intervention period with evaluations before, during, and after the intervention
* Have BP, HR, affective responses, and RPE measured at multiple time points
* Have EF, HRV, and salivary concentrations of NO biomarkers assessed before and after the intervention

DETAILED DESCRIPTION:
Physical training has been recommended as a non-pharmacological therapeutic strategy that can promote improvements in blood pressure levels in patients with systemic arterial hypertension (SAH). Resistance training (RT) has emerged due to the various benefits it promotes, including reducing blood pressure (BP) in this population, as improvements in heart rate variability (HRV) and endothelial function (EF). Guidelines suggest an intensity between 50% and 80% of 1 repetition maximum (1RM) in RT, reflecting a range of maximum repetitions between 9 and 26. However, there is a lack of studies that have made a direct comparison of the effect of different intensities in cardiovascular parameters of these patients. Therefore, the objective of this study will be to evaluate, acutely and chronically, the effect of RT intensity on BP, heart rate (HR), HRV, endothelial function, salivary concentrations of nitric oxide (NO) biomarker synthesis, also affectivity and rate of perceived exertion (RPE) of postmenopausal women with SAH. The study will be conducted in two stages, with two experiments: one acute and one chronic. In the acute experiment, with a crossover design, participants will perform the same RT session (with the order of these sessions being random), but in one condition they will train with 60% of 1RM and in another with 80% of 1RM. BP, HR and HRV will be measured before, at the end and for one hour after the session (hypotensive effect of the exercise). Affectivity will be measured before each test and at the end together with PSE. In the chronic study, participants will be randomized to one group that will train with 60% of 1RM and another group that will train with 80% of 1RM. Before, during and after the intervention, which will last 10 weeks, participants will be evaluated for BP, HR, affective responses and RPE, with EF, HRV and salivary concentrations of NO biomarkers measured before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Women with 50 to 65 old years;
* Postmenopausal diagnosis (amenorrhea for 12 months or more);
* Previous diagnosis of hypertension and treat with medications;
* Physically inactive.

Exclusion Criteria:

* History of other cardiovascular problems (heart failure, heart attack, stroke, etc);
* Grade II obesity (BMI ≥ 35 kg/m²);
* Medications (beta-blockers and/or non-dihydropyridine calcium channel blockers);
* Systolic blood pressure at rest above 160 mmHg and/or dyastolic blood presure above 105 mmHg;
* Unable to perform resistance exercise due to musculoskeletal or cognitive reasons.

Ages: 50 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-07-23 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Values of systolic and diastolic blood pressure (mmHg) | Up to end of study data collection (both stages), i.e, assesed up to 1 year
  This measurement will be assessed in both stages.
  In the acute phase, this measurement will be performed on the participant before, after and up to one hour after the end of the training session.
  In the chronic phase, this measure will be performed in participant after a rest in a quiet room with temperature controlled before (baseline) and after 10 week of intervention. Futhermore, along the intervention these measure will be performed before and after training sessions.

SECONDARY OUTCOMES:
Values of heart rate variability (ms) | Up to end of study data collection (both stages), i.e, assesed up to 1 year
  This measurement will be assessed in both stages.
  In the acute phase, this measurement will be performed on the participant before, after and up to one hour after the end of the training session.
  In the chronic phase, this measure will be performed in participant after a rest in a quiet room with temperature controlled before (baseline) and after 10 week of intervention. Futhermore, along the intervention these measure will be performed before and after training sessions.
Endothelial function (Flow mediated dilatation %) | Up to end of chronic experiment (baseline and post-intervention values), assesed up to 1 year
  This measurement will be performed before acute experiment (baseline) and after 10 week intervention (end of chronic experiment) in a quiet room with controlled temperature.
Salivary concentrations of nitric oxide (mmol/L) | Up to end of chronic experiment (baseline and post-intervention values), i.e, assesed up to 1 year
  This measurement will be performed before acute experiment (baseline) and after 10 week intervention (end of chronic experiment).
Rate of perceived exertion (scale from 1 to 10) | Up to end of study data collection (both stages), i.e, assesed up to 1 year
  This measurement will be performed after all training sessions, i.e, in both stages. The participants will be remembered the meanings of the scale.
Affectivity (scale from -5 to +5) | Up to end of study data collection (both stages), i.e, assesed up to 1 year
  This measurement will be performed before and after all training sessions, i.e, in both stages. The participants will be remembered the meanings of the scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Laboratório de Fisiologia do Exercício e Metabolismo, Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No